CLINICAL TRIAL: NCT03570515
Title: Yoga vs. Education for Restless Legs Syndrome - a Feasibility Study
Brief Title: Yoga vs. Education for Restless Legs Syndrome: a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1505699758
Record Dates: First submitted 2017-02-01; First posted 2018-06-27 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Yoga

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga (Experimental): Yoga group participants will attend two, 75-minute yoga classes/week for 4 weeks, then one class/week for 8 weeks, and do a 30-minute home practice on non-class days.
  Interventions: Behavioral: Yoga
- Educational Film (Active Comparator): Educational film group participants will attend one, 75-minute film class/week for 12 weeks, recording any RLS treatments they use at home.
  Interventions: Behavioral: Educational film

INTERVENTIONS:
Behavioral: Yoga — Yoga group participants will attend two, 75-minute yoga classes/week for 4 weeks, then one class/week for 8 weeks, and do a 30-minute home practice on non-class days, recording their practice on a yoga homework log provided to them.
  Arms: Yoga
Behavioral: Educational film — Educational film group participants will attend one, 75-minute film class/week for 12 weeks, recording any RLS treatments they use at home.
  Arms: Educational Film

SUMMARY:
The purpose of this study is to see whether adults with Restless Legs Syndrome (RLS) are willing to be in a 12-week study where they have a 50-50 chance of being placed in either a gentle yoga program or a film-based education program designed for people with RLS. If so, do they complete the program, and does their RLS, sleep, mood, or quality of life improve?

ELIGIBILITY:
Inclusion Criteria:

* ambulatory adults
* at least 21 years of age
* moderate-severe RLS, defined as:

  1. symptoms that meet all five of the International RLS Study Group essential diagnostic criteria for RLS (i.e., 1) an urge to move the legs, often associated with discomfort or disagreeable sensations in the legs, that 2) begins or worsen during periods of rest or inactivity; 3) is partially or totally relieved by movement; 4) is worse or only occurs in the evening or night; and 5) is not solely accounted for by another condition (e.g. leg cramps, positional discomfort, habitual foot tapping));
  2. RLS symptoms at least 1x/wk for the previous 3 months;
  3. a score of at least 2 points (moderate) IRLS question 6: "How severe was your RLS as a whole?"; and
  4. RLS diagnostic criteria applied as per training by the study physician, a sleep medicine expert; these criteria will help ensure exclusion of mimics (e.g. leg cramps, positional discomfort).
* willingness and ability to complete the 12-week yoga or educational film program and all study assessments;
* willingness to avoid use of any new drugs or treatments other than the assigned intervention.

Exclusion Criteria:

* practiced yoga within the past year;
* currently on dopaminergic agents (eg, ropinirole, pramipexole) or anti-psychotic medication;
* changed dosage if any other central nervous system agents (e.g., sedative hypnotics, gamma-aminobutyric acid (GABA) analogs, narcotic analgesics, antiadrenergic agents, or anticonvulsants) within the past 3 months;
* any orthopedic, neurologic or other condition that might prevent safe completion of a 12-week yoga program or confound assessments (e.g., neuropathy; Parkinson's disease; stroke; rheumatoid arthritis; renal failure; uncontrolled sleep apnea; recent (within the last 6 months) myocardial infarction; heart failure; cancer (other than non-melanoma skin cancer);
* pregnant or within 6 months post-partum).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-02-15 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 12 weeks
  To determine feasibility and acceptability of the programs, we will collect comprehensive information, both overall and by treatment group, on: rates of recruitment and success of different recruitment strategies, and reasons for refusal to participate.
Retention rates | 12 weeks
  To determine feasibility and acceptability of the programs, we will collect comprehensive information, both overall and by treatment group, on: rates of retention (completion of assessment visits)
Adherence rates | 12 weeks
  To determine feasibility and acceptability of the programs, we will collect comprehensive information, both overall and by treatment group, on rates of adherence (completion of home logs and class attendance rates (yoga and film groups); completion of home practice (yoga group));
Participant satisfaction | 12 weeks
  To determine feasibility and acceptability of the programs, we will collect comprehensive information, both overall and by treatment group, on participant satisfaction, assessed via a structured program evaluation questionnaire regarding participant perceptions of and experiences with the study, and satisfaction regarding their respective programs

SECONDARY OUTCOMES:
Yoga dosing preference | 12 weeks
  A structured questionnaire regarding possible yoga dosing scenarios will be administered at week 12 to determine participant preferences relative to yoga programs of varying duration and intensity (8 weeks, 16 classes (2x/week); 12 weeks, 16 classes (2x/week for the first 4 weeks, once/week thereafter); 16 weeks, 16 classes (once/week), as well as time of year the classes meet. Information from this questionnaire will aid in optimizing the yoga protocol for our future studies.
International RLS Rating Scale (IRLS) | 12 weeks
  To determine effect sizes of the programs, data critical to the design of the planned larger randomized clinical trial. RLS symptom severity, the primary efficacy outcome for the full scale trial, will be evaluated using the IRLS, a 10 item scale which includes questions related to frequency, intensity, and impact.
Pittsburgh Sleep Quality Index (PSQI) | 12 weeks
  Sleep quality will be assessed using the 9-item PSQI
Profile of Mood States (POMS) | 12 weeks
  Mood will be evaluated using the 65-item POMS
Perceived Stress Scale (PSS) | 12 weeks
  10-item PSS
Medical Outcomes Study Short Form-36 (SF-36). | 12 weeks
  Health-related quality of life will be measured using the 36-item SF-36.

CONTACTS AND LOCATIONS:
Overall Officials: Kim E Innes, PhD, Principal Investigator — WVU
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Selfe TK, Montgomery C, Klatt M, Wen S, Sherman KJ, Innes KE. An Exploratory Randomized Controlled Trial of a 12-Week Yoga Versus Educational Film Program for the Management of Restless Legs Syndrome: Feasibility and Acceptability. J Integr Complement Med. 2022 Apr;28(4):309-319. doi: 10.1089/jicm.2021.0182. Epub 2022 Jan 18. PMID 35426733
- [Derived] Innes KE, Selfe TK, Montgomery C, Hollingshead N, Huysmans Z, Srinivasan R, Wen S, Hausmann MJ, Sherman K, Klatt M. Effects of a 12-week yoga versus a 12-week educational film intervention on symptoms of restless legs syndrome and related outcomes: an exploratory randomized controlled trial. J Clin Sleep Med. 2020 Jan 15;16(1):107-119. doi: 10.5664/jcsm.8134. PMID 31957638
- [Derived] Selfe TK, Wen S, Sherman K, Klatt M, Innes KE. Acceptability and feasibility of a 12-week yoga vs. educational film program for the management of restless legs syndrome (RLS): study protocol for a randomized controlled trial. Trials. 2019 Feb 15;20(1):134. doi: 10.1186/s13063-019-3217-7. PMID 30770767